CLINICAL TRIAL: NCT06289608
Title: Bruxism and Underlying Psichological Factors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, JAVIER MONTERO, Full Professor, University of Salamanca
Other Study IDs: ID_2024
Record Dates: First submitted 2024-02-21; First posted 2024-03-04 (Actual); Last update posted 2024-03-04 (Actual); Status verified 2023-02

CONDITIONS: Bruxism; Muscular Disorders, Atrophic; Temporomandibular Joint Disorders
MeSH Terms: conditions — Bruxism; Muscular Disorders, Atrophic; Temporomandibular Joint Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Self-reported Bruxism: Those dental patients responding positively to at least 2 of the 6 items of the Pintado et al Self-reported Bruxism Inventory
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No dental intervention was made. Only a clinical examination

SUMMARY:
The aim of this study was o determine the relationship between self-reported bruxism (SB) and some psychological factors (i.e: Anxiety State-Trait; Stress Reactivity Index, Beck Depression Inventory). A consecutive sample of 101 patients that reported at least 2 of the 6 items of Bruxism self-reported index, were explored clinically for quantifying the number and severity of worn teeth, and also the severe and location of the muscular pain according to an standardized inventory.

DETAILED DESCRIPTION:
The Bruxism Self-Reported Index was that reported by Pintado et al.

Pintado MR, Anderson GC, DeLong R, Douglas WH. Variation in tooth wear in young adults over a two-year period. J Prosthet Dent. 1997;77:313-320.

The muscular pain was assessed by the last version of the Research Diagnostic Criteria reported by the Schiffman et al in 2014

Schiffman E, et al ; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Group†. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported Bruxism

Exclusion Criteria:

* Refused patients

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Self-reported bruxists
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Depression Level | baseline
  Beck Depression Index. The score range between 0-63, being proprotional to the current depression level
Stress Level | baseline
  Stress Reactitivy Index: Each of the 32 items are coded in a 4-point likert scale format, being 4 the worst category. The summary score is a proportional estimation of the stress level and range from 0-0.5 (minor stress), 0.6-1 (moderate stress) and >1 (severe stress)
Anxiety | baseline
  State-Trait Inventory has two estimation of anxiety, as a trait (assessed by 26 items) and as a transitory state (assessed by 20 items). All the items are coded in a 0-3 likert scale. The total score is proportional to the anxiety, being the threshold for determining anxiety above 20 points in male and 25 in females.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Odontológica de la Universidad de Salamanca, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No
The aggregated data will be published in a paper of the JCR Dentistry group